CLINICAL TRIAL: NCT02174146
Title: Effect of Non-surgical Periodontal Therapy on Leptin and Visfatin Expression in Gingival Tissues of Chronic Periodontitis With and Without Type 2 Diabetes Mellitus: A Study Utilizing ELISA and Real Time PCR
Brief Title: Leptin and Visfatin in Diabetic Patients With Periodontitis Before and After Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Ayman Ghallab, Associate Professor of periodontology, faculty of oral and dental medicine, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: leptin_visfatin_diabetes
Record Dates: First submitted 2014-06-23; First posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes Mellitus
Keywords: leptin; visfatin; chronic periodontitis; diabetes mellitus; non-surgical periodontal therapy
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- non-surgical therapy (Other): non-surgical periodontal therapy with ultrasonic scalers and periodontal curettes
  Interventions: Procedure: non-surgical periodontal therapy

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — supra and subgingival debridement
  Other Names: scaling and root planing

SUMMARY:
1. Are adipokines involved in pathogenesis of periodontal disease in diabetic patients?
2. Does their level change after periodontal therapy?

DETAILED DESCRIPTION:
Patients with chronic periodontitis only and patients with chronic periodontitis and diabetes were evaluated for levels of leptin and visfatin in the gingival tissues before and after non-surgical periodontal therapy.

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients having diabetes mellitus ≥5 years prior to the study.
* chronic periodontitis with clinical attachment loss > 5 mm.
* otherwise systemically healthy subjects.

Exclusion Criteria:

* any known systemic diseases other than diabetes.
* pregnancy or lactation.
* smokers.
* receiving periodontal treatment in the last 6 months.
* taking any drugs or medications other than anti-diabetic drugs.

Ages: 35 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
visfatin levels in gingival tissues | 3 months
  estimation of protein and gene expression of visfatin in patients with chronic periodontitis only and diabetic patients with periodontitis before and after non-surgical periodontal therapy..
leptin levels in gingival tissue | 3 months
  estimation of protein and gene expression of leptin in patients with chronic periodontitis only and diabetic patients with periodontitis before and after non-surgical periodontal therapy..

SECONDARY OUTCOMES:
pocket depth | 3 months
  estimation of pocket depth in patients with chronic periodontitis only and diabetic patients with periodontitis before and after non-surgical periodontal therapy.
clinical attachment level | 3 months
  estimation of clinical attachment level in patients with chronic periodontitis only and diabetic patients with periodontitis before and after non-surgical periodontal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Ghallab, M.D., Principal Investigator — Associate Professor of periodontology faulty of oral and dental medicine Cairo Unv.
Locations (1):
- Faculty of oral and dental medicine, Cairo, Egypt

REFERENCES:
- [Result] Pradeep AR, Raghavendra NM, Sharma A, Patel SP, Raju A, Kathariya R, Rao NS, Naik SB. Association of serum and crevicular visfatin levels in periodontal health and disease with type 2 diabetes mellitus. J Periodontol. 2012 May;83(5):629-34. doi: 10.1902/jop.2011.110272. Epub 2011 Oct 3. PMID 21966944
- [Result] Pradeep AR, Raghavendra NM, Prasad MV, Kathariya R, Patel SP, Sharma A. Gingival crevicular fluid and serum visfatin concentration: their relationship in periodontal health and disease. J Periodontol. 2011 Sep;82(9):1314-9. doi: 10.1902/jop.2011.100690. Epub 2011 Feb 10. PMID 21309715
- [Result] Raghavendra NM, Pradeep AR, Kathariya R, Sharma A, Rao NS, Naik SB. Effect of non surgical periodontal therapy on gingival crevicular fluid and serum visfatin concentration in periodontal health and disease. Dis Markers. 2012;32(6):383-8. doi: 10.3233/DMA-2012-0897. PMID 22684235
- [Result] Karthikeyan BV, Pradeep AR. Leptin levels in gingival crevicular fluid in periodontal health and disease. J Periodontal Res. 2007 Aug;42(4):300-4. doi: 10.1111/j.1600-0765.2006.00948.x. PMID 17559625
- [Result] Karthikeyan BV, Pradeep AR. Gingival crevicular fluid and serum leptin: their relationship to periodontal health and disease. J Clin Periodontol. 2007 Jun;34(6):467-72. doi: 10.1111/j.1600-051X.2007.01078.x. Epub 2007 Apr 23. PMID 17451417
- [Result] Johnson RB, Serio FG. Leptin within healthy and diseased human gingiva. J Periodontol. 2001 Sep;72(9):1254-7. doi: 10.1902/jop.2000.72.9.1254. PMID 11577959
- [Result] Bozkurt FY, Yetkin Ay Z, Sutcu R, Delibas N, Demirel R. Gingival crevicular fluid leptin levels in periodontitis patients with long-term and heavy smoking. J Periodontol. 2006 Apr;77(4):634-40. doi: 10.1902/jop.2006.050277. PMID 16584344